CLINICAL TRIAL: NCT06265610
Title: A Comparison Of The Effect Of Target-Controlled Infusion Anesthesia And Inhalation Anesthesia On Patient Outcomes In Pediatric Patients Undergoing Endovascular Intervention
Brief Title: A Comparison Of The Effect Of Target-Controlled Infusion Anesthesia And Inhalation Anesthesia
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sibel Seçkin Pehlivan, Principal Investigator, TC Erciyes University
Other Study IDs: 2022/186
Record Dates: First submitted 2024-01-12; First posted 2024-02-20 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Patients; Cardiology
Keywords: Sevoflurane,; Propofol; Target Controlled Infusion,

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: Total intravenous anesthesia with target-controlled infusion (TCI/TIVA) was applied as an anesthesia method to be applied to patients during cardiology angiography procedures.
  Interventions: Procedure: TIVA/TCI
- Group 2: In the anesthesia method to be applied to patients during cardiology angiography procedures, inhalation anesthesia was applied.

INTERVENTIONS:
Procedure: TIVA/TCI — : The aim of this study was to evaluate the effects of total intravenous anesthesia with target-controlled infusion (TCI/TIVA) on intraoperative hemodynamic parameters and postoperative awakening criteria in pediatric endovascular intervention patients
  Other Names: Inhalatıon
  Groups: group 1

SUMMARY:
A total of 70 patients who underwent angiographic examination, ASD closure, VSD closure, PDA closure and aortic balloon dilatation were included in this study.

DETAILED DESCRIPTION:
A total of 70 patients who underwent angiographic examination, ASD closure, VSD closure, PDA closure and aortic balloon dilatation were included in this study. Patients underwent standard electrocardiography (ECG) monitoring with heart rate (HR), noninvasive blood pressure (NIKB), peripheral oxygen saturation (SpO2) and Bispectral index (BIS). Baseline NIKB, SpO2 and HR were recorded before the procedure, intraoperatively and in the postoperative recovery unit. In the postoperative recovery unit, the patient's recovery time was also evaluated and recorded with the Modified Aldrete Recovery Score.

ELIGIBILITY:
Inclusion Criteria:

1. Children weighing over 10 kg and between the ages of 3-18 who will undergo angiography
2. Patients who are not allergic to the drugs used

Exclusion Criteria:

1. ASA Ⅳ patients
2. Patients with Diabetes Mellitus
3. Patients with severe lung disease
4. Patients with psychiatric disorders
5. Patients with opioid addiction -

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children ages 3 to 18 with heart disease
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
intraoperative period | an average of 2 hours
  During cardiology angiography procedures, patients' heart rate,measurements will be evaluated.
postoperative period | an average of 2 hours
  During cardiology angiography procedures, patients' eye opening time will be evaluated.
hemodynamic parameters | an average of 2 hours
  During cardiology angiography procedures, patienheart ts' mean arterial pressure (MAP),measurements will be evaluated.

SECONDARY OUTCOMES:
Modified Aldrete Recovery Score | during the processing period
  Modified Aldrete Recovery Score will be evaluated in the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Pehlivan, MD, Study Director — TC Erciyes University; Mustafa Cakıllı, Principal Investigator — Department of Anaesthesiology and Reanimation, Yozgat City Hospital,; Ozlem OZ GERGIN, MD, Principal Investigator — Department of Anaesthesiology and Reanimation, Medical Faculty, Erciyes University; Ali BAYKAN, Prof, Principal Investigator — Department of Pedıatrıc Cardiology, Medical Faculty, Erciyes University; Recep AKSU, Prof, Principal Investigator — Department of Anaesthesiology and Reanimation, Medical Faculty, Erciyes University; Karamehmet YILDIZ, prof, Principal Investigator — Department of Anaesthesiology and Reanimation, Medical Faculty, Erciyes University
Locations (1):
- Sibel Seçkin Pehlivan, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared upon reasonable request to the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data can be shared upon reasonable request to the corresponding author.
Access Criteria: Data can be shared upon reasonable request to the corresponding author.

REFERENCES:
- [Result] Lerman J, Johr M. Inhalational anesthesia vs total intravenous anesthesia (TIVA) for pediatric anesthesia. Paediatr Anaesth. 2009 May;19(5):521-34. doi: 10.1111/j.1460-9592.2009.02962.x. No abstract available. PMID 19453585
- [Result] Lerman J. TIVA, TCI, and pediatrics: where are we and where are we going? Paediatr Anaesth. 2010 Mar;20(3):273-8. doi: 10.1111/j.1460-9592.2009.03238.x. Epub 2010 Jan 19. PMID 20102520